CLINICAL TRIAL: NCT05390190
Title: Non Ablative Radiofrequency in the Treatment of Onychomycosis, a Pilot Study
Brief Title: Radiofrequency in Onychomycosis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Hagar El Sayed, Dr, Cairo University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: onychomycosis
Record Dates: First submitted 2022-05-20; First posted 2022-05-25 (Actual); Last update posted 2022-05-25 (Actual); Status verified 2022-05

CONDITIONS: Onychomycosis
MeSH Terms: conditions — Onychomycosis

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Non ablative radiofrequency (Experimental): Device
  Interventions: Device: Non ablative radiofrequency

INTERVENTIONS:
Device: Non ablative radiofrequency — Device

SUMMARY:
Onychomycosis is the most common nail disease, representing more than 50% of all onychopathies.

DETAILED DESCRIPTION:
Treatments with antifungals may not be successful due to several factors, including the long time required to apply topical medications, the side effects of systemic drugs, and the application of insufficient medication to the target area. Non-ablative radiofrequency devices can be used to treat onychomycosis without harming the nail matrix cells.

ELIGIBILITY:
Inclusion Criteria:

* Onychomycosis patients

Exclusion Criteria:

Patients with excessive manual work

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 20 (Estimated)
Dates: Start 2022-07-01 (Estimated); Primary Completion 2022-10-01 (Estimated); Study Completion 2022-10-01 (Estimated)

PRIMARY OUTCOMES:
Onychomycosis severity index | 3 months
  Clinical assessment